CLINICAL TRIAL: NCT02157298
Title: A 16-week Multicenter, Randomized, Parallel-group, Double-blind, Placebo-controlled Phase IV Study With a 36-week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin Therapy When Added to the Therapy of Japanese Patients With Type 2 Diabetes With Inadequate Glycemic Control on Insulin
Brief Title: Phase IV Study With a 36-week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin Therapy When Added to the Therapy of Japanese Patients With Type 2 Diabetes With Inadequate Glycemic Control on Insulin.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1692C00013
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Japanese patients with type 2 diabetes with inadequate glycemic control on insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dapagliflozin 5mg (Experimental): dapagliflozin tablet 5mg
  Interventions: Drug: Dapagliflozin 5 mg
- Placebo (Placebo Comparator): dapagliflozin tablet 5mg placebo
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Dapagliflozin 5 mg — Dapagliflozin, a blood glucose lowering drug. Oral dose
  Arms: dapagliflozin 5mg
Drug: Placebo tablet — Placebo tablet. Oral dose
  Arms: Placebo

SUMMARY:
Japanese male and female patients with Type 2 Diabetes and aged ≥ 20 years old, with inadequate glycemic control on insulin defined as Haemoglobin A1c ≥ 7.2% and < 11% will be enrolled into the wash-out phase or directly into the lead-in phase depending on whether the patient has been receiving an Oral antidiabetic drug (including Glucagon-Like Peptide-1 agonists and excluding Thiazolidinedions) other than a Dipeptidyl Peptidase-4 inhibitor as part of the baseline treatment. Additional treatment with a concomitant Dipeptidyl Peptidase-4 inhibitor is allowed. And around 180 eligible patients in total will be randomized into the study with a 2:1 randomization scheme (i.e.120 patients into the dapagliflozin treatment group and 60 patients into the placebo treatment group. All subjects who completed a 16 weeks double-blind treatment period will shift to a 36 weeks open extension treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of Type 2 Diabetes according the criteria specified by the Japan Diabetes Society
* Japanese Men or women age ≥ 20 years at time of consenting.
* Stable (unless adjustment is required based on Fasting Plasma Glucose values) dose insulin* mono-therapy with the mean insulin [up to two types of insulin within authorized indication in Japan] dose of ≥ 0.2 IU/kg/day AND ≥ 15 IU/body/day over the past 8 weeks prior to enrolment.
* HbA1c ≥ 7.2% and < 11% from the blood samples collected at Visit 1 (enrolment) and Visit 3, observed from the central laboratory

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus, known diagnosis of Maturity Onset Diabetes of the Young, secondary diabetes mellitus or diabetes insipidus
* History of diabetic ketoacidosis.
* Thyroid-stimulating hormone and free T4 values outside normal range, observed from the central laboratory; an abnormal Thyroid-stimulating hormone value needs to be followed up with a free T4 test. Patients with abnormal free T4 values will be excluded at Visit 1
* Fasting Plasma Glucose >240 mg/dL (twice in a row) despite the permitted dose adjustment of insulin therapy during washout period and lead-in period.
* Recent cardiovascular events in a patient.
* eGFR <45 mL/min/1.73 m2 at Visit 3, observed from the central laboratory.
* History of unstable or rapidly progressing renal disease.
* History of unexplained microscopic or gross hematuria, or microscopic hematuria at Visit 1, confirmed by a follow-up sample at next scheduled visit, where according to the investigator a satisfactory evaluation of hematuria has not been conducted.
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN, observed from the central laboratory at Visit 1.
* Total bilirubin >2.0 mg/dL (34.2 μmol/L), observed from the central laboratory at Visit 1.
* Positive serologic evidence of current infectious liver disease including Hepatitis A viral antibody IgM, Hepatitis B surface antigen and Hepatitis C virus antibody, observed from the central laboratory.
* Haemoglobin <10 g/dL (<100 g/L) or 6.2 mmol/L for men; haemoglobin <9.0 g/dL (<90 g/L) or 5.9 mmol/L for women, observed from the central laboratory at Visit 1.
* History of chronic haemolytic anaemia or haemoglobinopathies (for example, sickle cell anaemia, thalassemia, sideroblastic anaemia). Mild haemolysis due to artificial heart valves or due to sickle cell trait is not an exclusion criterion except when haemoglobin levels are too low (as defined in haemoglobin criteria above).
* History of malignancy within the last 5 years prior to enrolment, excluding successful treatment of basal or squamous cell skin cancer.

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Research Site, Adachi-ku
  - Research Site, Chitose-shi
  - Research Site, Chiyoda-ku
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Kamakura-shi
  - Research Site, Koriyama-shi
  - Research Site, Mitaka-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sendai
  - Research Site, Shizuoka
  - Research Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 06-Jun-2014; Last participant last visit of ST period: 02-Feb-2015; 266 participants were enrolled in 20 Japanese centers. 183 Japanese men or women aged >=20 years with inadequate glycemic control (HbA1c levels of >=7.2% to <11.0%) with diet, exercise and on stable dose of insulin +/- DPP-4 inhibitor were treated.
Pre-assignment Details: A 8-week wash-out period was applicable only for participants on ongoing anti-diabetic treatment at enrollment. A 2-week lead-in period was applicable for all participants.
Groups:
- Dapagliflozin: Dapagliflozin 5 mg plus insulin alone or in combination with DPP-4 inhibitor
- Placebo: Placebo plus insulin alone or in combination with DPP-4 inhibitor
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 123 | 60
Completed | 119 | 58
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Subject no longer meets study criteria | 1 | 2
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during the short-term double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 122 | 60 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.83) | 57.6 (9.86) | 58.0 (9.82)
Age, Customized [Number; unit: participants]
  <=65 years | 84 | 43 | 127
  Between 65 and 75 years | 37 | 16 | 53
  >=75 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 89 | 40 | 129
Region of Enrollment [Number; unit: participants]
  Japan | 122 | 60 | 182
Body Weight [Mean (Standard Deviation); unit: kg] | 73.90 (15.663) | 71.89 (13.430) | 73.24 (14.956)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.89 (4.930) | 26.12 (3.485) | 26.64 (4.510)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 93.2 (11.83) | 92.3 (9.00) | 92.9 (10.96)
HbA1c [Mean (Standard Deviation); unit: percent of hemoglobin glycosylated] | 8.26 (0.792) | 8.52 (0.937) | 8.34 (0.849)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 160.70 (44.948) | 159.68 (38.001) | 160.36 (42.679)
Calculated Mean Daily Insulin Dose [Mean (Standard Deviation); unit: IU/Day] | 37.87 (18.033) | 40.58 (16.764) | 38.76 (17.625)
DPP-4 Inhibitor Usage [Number; unit: participants]
  Yes | 54 | 27 | 81
  No | 68 | 33 | 101

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: Mean change in HbA1c levels from baseline to Week 16 between dapagliflozin 5 mg versus placebo
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and at least one post-baseline value up to week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hemoglobin glycosylated
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 122 | 59
percentage of hemoglobin glycosylated | -0.55 [-0.67 to -0.42] | 0.05 [-0.13 to 0.23]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(dapa) minus mean(placebo) = 0 versus alternative HA: mean(dapa) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significant at alpha=0.05 (two-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure; with fixed categorical effects of treatment, week, DPP-4, baseline eGFR, treatment-by-week interaction, continuous fixed covariate of baseline value; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.81 to -0.39], Standard Error of Mean 0.1053

2. Secondary Outcome: Fasting Plasma Glucose
Description: Mean change in fasting plasma glucose from baseline to Week 16 between dapagliflozin 5 mg versus placebo
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and at least one post-baseline value up to week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 121 | 59
mg/dL | -21.7 [-28.3 to -15.1] | 1.0 [-8.4 to 10.3]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(dapa) minus mean(placebo) = 0 versus alternative HA: mean(dapa) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-33.2 to -12.2], Standard Error of Mean 5.301

3. Secondary Outcome: Total Body Weight
Description: Mean change in total body weight from baseline to Week 16 between dapagliflozin 5 mg versus placebo
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and at least one post-baseline value up to week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 122 | 59
kg | -0.6 [-0.9 to -0.2] | 0.7 [0.2 to 1.1]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(dapa) minus mean(placebo) = 0 versus alternative HA: mean(dapa) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.7 to -0.7], Standard Error of Mean 0.255

4. Secondary Outcome: Total Mean Daily Insulin Dose
Description: Mean change in calculated mean daily insulin dose from baseline to Week 16 between dapagliflozin 5 mg versus placebo
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and at least one post-baseline value up to week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/Day
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 121 | 60
IU/Day | -0.74 [-1.21 to -0.27] | -0.02 [-0.68 to 0.64]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(dapa) minus mean(placebo) = 0 versus alternative HA: mean(dapa) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0743, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.51 to 0.07], Standard Error of Mean 0.4017

5. Secondary Outcome: Proportion of Participants With Mean Daily Insulin Dose Reduction of Greater Than or Equal 10%
Description: Proportion of participants with mean daily insulin dose reduction greater than or equal 10% from baseline to week 16 (LOCF) between dapagliflozin 5 mg versus placebo
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and Week 16 (LOCF) value
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 121 | 60
percentage of participants | 8.2 [3.3 to 13.1] | 4.9 [-0.7 to 10.4]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: proportion(dapa) minus proportion(placebo) = 0 versus alternative HA: proportion(dapa) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.3727, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Tsitatis, Davidian, Zhang & Lu, with adjustment with adjustment for baseline value and DPP-4; Risk Difference (RD) = 3.4, 95% CI 2-sided [-4.0 to 10.7], Standard Error of Mean 3.769

ADVERSE EVENTS:
Time Frame: Non-serious/serious adverse events on or after the first date of double-blind treatment and on or prior to the last day plus 4/30 days or up to follow-up visit if earlier, or up to and excluding the start date of open-label extension period if earlier.
Description: Participants were questioned at each study about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/123 | 0/60
Other Adverse Events (participants affected / at risk) | 24/123 | 10/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=123) | Placebo (N=60)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=123) | Placebo (N=60)
Nasopharyngitis (Infections and infestations) | 13 | 7
Pollakiuria (Renal and urinary disorders) | 11 | 3
Constipation (Gastrointestinal disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
For HbA1c, FPG and TBW: excluding data after insulin up-titration and for Mean Daily Insulin Dose: including data after insulin up-titration were used. For participants who did not complete week 16 last observation carried forward (LOCF) was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.